CLINICAL TRIAL: NCT02981576
Title: Comparative Evaluation of Safety and Effectiveness of Autologous Bone Marrow Derived Mesenchymal Stem Cells (BM-MSC) vs Adipose Tissue Derived Mesenchymal Stem Cells (AT-MSC) in the Treatment of Spinal Cord Injury (SCI) Patient.
Brief Title: Safety and Effectiveness of BM-MSC vs AT-MSC in the Treatment of SCI Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCIUJCTC
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Mesenchymal Stem Cells
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recipient of AT-MSC (Active Comparator): Patients who will receive Autologous Mesenchymal Stem Cells from AdiposeTissue by Intrathecal injection of stem cells that will be performed 3 times.
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- Recipient of BM-MSC (Active Comparator): Patients who will receive Autologous Mesenchymal Stem Cells from Bone marrow by Intrathecal injection of stem cells that will be performed 3 times.
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — Autologous Mesenchymal Stem Cells will be collected from patients, prepared in the lab and then injected intrathecally.

SUMMARY:
Spinal Cord Injury (SCI) is a devastating condition that leads to permanent functional and neurological deficits in injured individuals. The limited ability of the Central Nervous System (CNS) to spontaneously regenerate impairs axonal regeneration and functional recovery of the spinal cord. The leading causes are motor-vehicle crashes, sports-associated accidents, falls, and violence-related injuries.

Unfortunately, there is still no effective clinical treatment for SCI. In recent years, tissue engineering and regenerative medicine based approaches have been proposed as alternatives for SCI repair/regeneration. Mesnchymal stem cells (MSC) use in SCI showed promising results in several studies. Our aim is to assess and compare the safety and effectiveness of autologous BM-MSC vs autologous AT-MSC in these patients.

DETAILED DESCRIPTION:
The study will be conducted at Cell Therapy Center (CTC) in Jordan, where 14 SCI patients meeting the inclusion criteria will be recruited and blindly divided into 2 groups of equal numbers. The first groups will be treated with autologous BM-MSC, while the second group will be treated with autologous AT-MSC. The outcomes and improvements will be assessed using the American Spinal Injury Association (ASIA) Impairment Scale (AIS). Magnetic Resonance Imaging (MRI) will be performed at base line and after 12 months of the stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Complete spinal cord injury grade AIS-A or -B, or incomplete C
* At least 2 weeks since time of injury
* Cognitively unaffected
* Motivated for stem cell transplantation

Exclusion Criteria:

* Reduced cognition
* Age under 18 years of above 70 years
* Significant osteoporosis in spine and/or joints
* Pregnancy (Adequate contraceptive use is required for women in fertile age)
* Anoxic brain injury
* Neurodegenerative diseases
* Evidence of meningitis
* Positive serology for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Syphilis.
* Medical Complications that contraindicate surgery, including major respiratory complications.
* Use of metal implants close to vascular structures (such as cardiac pacemaker or prosthesis) that contraindicate Magnetic resonance imaging (MRI).
* Other medical conditions which can interfere with stem cell transplantation
* Inability to provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05-05 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Comparing the number of side effects and the improvement on ASIA Impairment score between SCI patients receiving autologous AT-MSC vs BM-MSC. | 12 months
  Comparing the number of SCI patients with any relevant side effects observed and the measured outcome in each arm by follow up Magnetic Resonance Imaging (MRI) and clinical signs and symptoms using ASIA scoring system..

SECONDARY OUTCOMES:
Investigating the number of side effects in SCI patients receiving autologous BM-MSC. | 12 months
  Assessing the number of SCI patients with any relevant side effects observed.
Investigating the effectiveness of autologous BM-MSC in treating SCI patients. | 12 months
  Assessing the therapeutic benefits of the injected Autologous BM-MSC by follow up Magnetic Resonance Imaging (MRI) and clinical signs and symptoms using ASIA scoring system.
Investigating the number of side effects in SCI patients receiving autologous AT-MSC. | 12 months
  Assessing the number of SCI patients with any relevant side effects observed.
Investigating the effectiveness of autologous AT-MSC in treating SCI patients. | 12 months
  Assessing the therapeutic benefits of the injected Autologous AT-MSC by follow up Magnetic Resonance Imaging (MRI) and clinical signs and symptoms using ASIA scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Awidi, MD, Study Chair — University of Jordan
Locations (1):
- Cell Therapy Center, University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cell Therapy Center Website — http://centers.ju.edu.jo/en/ctc/Home.aspx